CLINICAL TRIAL: NCT01314989
Title: Effect of Cyproheptadine on Weight Gain and Feeding Behavior in 2 to 4 Years Old Children With Failure to Thrive
Brief Title: Cyproheptadine as an Appetite Stimulant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Dr Valerie Marchand, Ste-Justine University Health Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Cypro-24
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Failure to Thrive
MeSH Terms: conditions — Failure to Thrive | interventions — Cyproheptadine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyproheptadine (Active Comparator): Cross-over study
  Interventions: Drug: Cyproheptadine
- Sugar pill (Placebo Comparator): Cross-over study
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Cyproheptadine — 0,25mg/kg/day orally in 2 doses per day (2mg/5 ml)for 1 month
  Arms: Cyproheptadine
Drug: Sugar pill — liquid placebo
  Arms: Sugar pill

SUMMARY:
Cyproheptadine is currently clinically used as an appetite stimulant for children with failure to thrive without underlying organic disease. Otherwise, no randomised control trial demonstrates the efficacy of Cyproheptadine on those patients. This is precisely what the investigators intend to demonstrate on this randomised placebo control cross-over trial. Our hypothesis is that Cyproheptadine is more efficient than placebo to improve weight gain and feeding behaviour on 2 to 4 years old children with failure to thrive.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 4 years of age
* failure to thrive

Exclusion Criteria:

* Medication affecting appetite
* Medication interacting with Cyproheptadine
* Prematurity under 36 weeks of gestation
* Neurologic impairment
* underlying organic disease

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-03 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Weight gain | January 2011 to January 2012

SECONDARY OUTCOMES:
Feeding behaviour | January 2011 to January 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Ste-Justine University Health Center, Montreal, Quebec, Canada